CLINICAL TRIAL: NCT07206615
Title: Post Market Clinical Follow-Up Study - Chart Review of the Spot Ex Endoscopic Marker
Brief Title: Spot Ex PMCF 01 Study
Acronym: Spot Ex PMCF
Status: Enrolling by invitation | Type: Observational
Sponsor: Laborie Medical Technologies Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN-00082
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Presence of Spot Ex Endoscopic Marker
Keywords: Spot Ex; Endoscopic Marker; Laborie

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | US Export: Yes

GROUPS / COHORTS (1):
- Spot Ex Endoscopic Marker: Subjects with Spot Ex Endoscopic Marker present 36 months post-tattoo
  Interventions: Other: Endoscopic marker

INTERVENTIONS:
Other: Endoscopic marker — Study to confirm the safety and performance of the Laborie Spot Ex Endoscopic Marker in accordance with the approved labelling/instructions for use (IFU).

SUMMARY:
Post market clinical study that is a chart review of the Spot Ex Endoscopic Marker

DETAILED DESCRIPTION:
This study is a medical chart review to confirm the safety and performance of the Spot Ex Endoscopic Marker in accordance with the approved labelling/instructions for use (IFU).

ELIGIBILITY:
Inclusion Criteria:

* Patients who had a marking in their GI tract with the Spot Ex Endoscopic marker for the purposes of clinical surveillance.

Exclusion Criteria:

* 1. Patients who had the marked tissue resected less than 3 years after initial marking.
* 2. Inadequate medical documentation to ascertain visualization of the marking.
* 3. Inability to visualize or image the marking due to poor colonoscopy preparation.
* 4. Patients considered as Vulnerable Populations, as defined in CFR - Code of Federal Regulations Title 21

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 subjects with visual confirmation of the presence of Spot Ex as visualized by a clinician or in colonoscopy imaging at 36 months. Additional subjects may be screened to reach the minimum sample size required (60 subjects).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Longevity | From endoscopic marker placement date to 36 months post-tattoo date
  Visual confirmation at 36 months - Percent of subjects with visual confirmation of the presence of Spot Ex as visualized by a clinician or in colonoscopy imaging at 36 months.

SECONDARY OUTCOMES:
Safety Endpoint | From endoscopic marker placement date to 36 months post-tattoo date
  Percent of treatment-related adverse events specified in the protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- IU Health University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided